CLINICAL TRIAL: NCT04702230
Title: Value of Functional Magnetic Resonance Imaging of Hepatocellular Carcinoma After Transarterial Chemoembolization or Transarterial Radioembolization
Status: Terminated | Type: Observational
Why Stopped: Treatment practice unexpectedly changed during the course of the study. Majority of follow-up MRI performed in external institutions. Consequently, the planned number of participants could not be reached.
Sponsor: University of Zurich (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Caecilia Reiner, Staff Radiologist, University of Zurich
Other Study IDs: BASEC ID 2016-01868
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Liver Neoplasm
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post-TAE
  Interventions: Diagnostic Test: MRI
- post-TARE
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Baseline and follow-up MRI at 1 and 3 months post-TAE or post-TARE

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common malignancies worldwide and is commonly treated with transarterial locoregional therapies (transarterial chemoembolization (TACE) or transarterial radioembolization (TARE)). Early assessment of the effectiveness of transarterial locoregional therapies is critical for treatment planning and early identification of non-responders to allow a timely repeat treatment or conversion to a second-line local-regional or systemic treatment. Response of HCC to transarterial locoregional therapies is usually assessed by changes in tumor contrast material enhancement thought to reflect tumor viability. However, contrast material enhancement may not always accurately indicate tumor response as it may also reflect reactive changes rather than residual tumor tissue. A potential alternative for evaluation of the residual tumor is diffusion-weighted imaging (DWI), which can differentiate between tumor tissue with high cellularity and tumor necrosis. DWI has been shown useful in therapy response assessment of liver tumors. A further development of DWI is intravoxel incoherent motion imaging (IVIM), an MRI technique which also takes tumor perfusion and thus tumor viability into account. This makes IVIM a promising tool for early therapy response assessment in HCC patients.

The primary objective is to proof that DWI and especially IVIM with its inherent perfusion information related to tumor neovascularization allows for reliable and quantitative monitoring of tumor response and separating responders from non-responders to either of the two locoregional treatments (TACE or TARE) The secondary objective is to identify whether DWI/IVIM acquired during early follow-up (1 month after treatment) leads to better response assessment than DWI/IVIM acquired during later follow-up (3 months after treatment).

The primary outcome will be the DWI/IVIM values in patients responding to transarterial locoregional therapies of HCC compared to patients not responding to therapy according to mRECIST at 6 months The secondary outcome will be the number of patients correctly identified as responders at early follow-up (after 1 month) with DWI/IVIM compared to the number of patients correctly identified as resopnders at later follow-up (after 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Male and Female patients ≥18 years of age
* Patients with HCC according to imaging findings and/or histology and scheduled for TACE or TARE

Exclusion Criteria:

* Women who are pregnant or breast feeding,
* Please note that female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study,
* Patients with impaired renal function (estimated glomerular filtration rate <30 ml/min)
* Patients with non-MRI compatible metallic or electronic implants, devices or metallic foreign bodies (cardiac pacemaker, shrapnel, cochlea implants, neurostimulator, or other non-MRI compatible implants).
* Tumor-directed therapy (i.e. systemic chemotherapy) between transarterial therapy and 3-months follow-up MRI exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with HCC according to imaging findings and/or histology and scheduled for TACE or TARE
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
DWI/IVIM values | 6 months
  DWI/IVIM values in patients responding to transarterial locoregional therapies of HCC compared to patients not responding to therapy according to mRECIST at 6 months

SECONDARY OUTCOMES:
early responders | 6 months
  The secondary outcome will be the number of patients correctly identified as responders at early follow-up (after 1 month) with DWI/IVIM compared to the number of patients correctly identified as resopnders at later follow-up (after 3 months).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No